CLINICAL TRIAL: NCT01544894
Title: Comparison of Raloxifene and Strontium Ranelate on Compliance and Efficacy in Women With Postmenopausal Osteoporosis
Brief Title: Clinical Study of Raloxifene and Strontium Ranelate in Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Antonio Cano Sanchez, Professor in Obstetrics and Gynecology, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sr-ral-postmOTP
Record Dates: First submitted 2012-01-18; First posted 2012-03-06 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Postmenopausal Osteoporosis; Compliance
Keywords: Postmenopausal osteoporosis; Compliance; Bone mineral density; Bonemarkers
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Patient Compliance | interventions — Raloxifene Hydrochloride; strontium ranelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- raloxifene (Active Comparator): 60 mg/d for one year.
  Interventions: Drug: Raloxifene
- strontium ranelate (Active Comparator): 2 g/d for one year.
  Interventions: Drug: Strontium ranelate

INTERVENTIONS:
Drug: Raloxifene — 60 mg/d for one year
  Other Names: Evista
  Arms: raloxifene
Drug: Strontium ranelate — 2 g/d, for one year
  Other Names: Protelos
  Arms: strontium ranelate

SUMMARY:
The purpose of this study was to compare compliance and efficacy of raloxifene and strontium ranelate in a group of women with postmenopausal osteoporosis.

DETAILED DESCRIPTION:
OBJECTIVE: To compare the performance of raloxifene and strontium rannelate in the management of women with postmenopausal osteoporosis.

DESIGN: Prospective, open label study. SETTING: University hospital menopause unit. PATIENTS: 80 women with postmenopausal osteoporosis were assigned to either raloxifene (60 mg/d) or strontium ranelate (2g/d). Participants were followed for 1 year.

MAIN OUTCOME MEASURE(S): Compliance with each regime. Secondary objectives were parameters of efficacy, including changes in bone mineral density and bone biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with densitometric osteoporosis

Exclusion Criteria:

* Secondary osteoporosis

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Clinical study of raloxifene and strontium ranelate in postmenopausal osteoporosis | One year
  Primary Outcome measure: compliance. Assessment of compliance assessed two variables, the number of participants maintaining treatment after one year and, among those that completed the one year treatment, the number of them that completed at least 80% of the prescribed dose.

SECONDARY OUTCOMES:
Clinical study of raloxifene and strontium ranelate in postmenopausal osteoporosis | One year
  Secondary outcome measure: efficacy. Efficacy has been assessed by changes in axial bone mineral density (spine and hip) and by changes in biochemical bone markers (C-telopeptides and P1NP in serum).
  Axial densitometry has been performed prior to treatment and after completion of the programmed one-year treatment.
  Bone markers have been assessed prior to treatment and at the 3rd, 6th and 12th month of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cano, MD, Study Director — University of Valencia
Locations (1):
- Hospital Universitario Dr Peset, Valencia, Valencia, Spain